CLINICAL TRIAL: NCT01283087
Title: Spinal Anesthesia Using Lidocaine and Sufentanil and TNS (=Transient Neurological Symptoms)
Brief Title: Spinal Anesthesia Using Lidocaine and Sufentanil and (Transient Neurological Symptoms) TNS
Status: Completed | Type: Observational
Sponsor: Vestre Viken Ringerike Sykehus (Other)
Responsible Party: Principal Investigator, Britt-Marie Berling, MD, PhD, Vestre Viken Ringerike Sykehus
Other Study IDs: 400229
Record Dates: First submitted 2011-01-21; First posted 2011-01-25 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Transient Neurologic Symptoms
Keywords: TNS; Spinal anesthesia; Lidocaine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to find out whether patients receiving spinal anesthesia containing lidocaine and sufentanil get transient neurological symptoms.

ELIGIBILITY:
Inclusion Criteria:

* adults over the age of seventeen years

Exclusion Criteria:

* patient refuse spinal anesthesia
* spinal anesthesia is contraindicated
* pregnancy
* patient is incapable of giving consent
* diabetes
* neurological disorders
* chronic pain
* chronic use of analgesics
* spinal anesthesia within five days before the actual surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are submitted for surgery at a local hospital and where spinal anesthesia is indicated.
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2011-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Symptoms of transient neurological symptoms | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: halfdan Aas, MD, PhD, Study Chair — Vestre Viken HF; halfdan Aas, MD, PhD, Study Chair — VestreViken HF
Locations (2):
- Norway (2):
  - Ringerike Sykehus, Hønefoss
  - Vestre Viken HF Ringerike Sykehus, Hønefoss